CLINICAL TRIAL: NCT01234155
Title: Exercise Training and Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Thomas Solomon, Group Leader, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-1-2010-027
Record Dates: First submitted 2010-11-01; First posted 2010-11-04 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2014-12

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Exercise; Diabetes; Obesity; Insulin Sensitivity; Insulin Secretion; Beta-cell Function; Glycemic Control; GIP; GLP-1
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Motor Activity; Diabetes Mellitus; Obesity; Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control (No Intervention)
- Exercise - Continuous Walking (Experimental)
  Interventions: Behavioral: Exercise - Continuous Walking
- Exercise - Interval Walking (Experimental)
  Interventions: Behavioral: Exercise Training - Interval Walking

INTERVENTIONS:
Behavioral: Exercise Training - Interval Walking — Duration: 4 months. Exercise training sessions will be performed 3-5 days/week. Sessions will consist of walking for 3 minutes at 70% VO2max followed by 3 minutes at 40% VO2max for up to 60 minutes/day.
  Arms: Exercise - Interval Walking
Behavioral: Exercise - Continuous Walking — Duration: 4 months. Exercise training sessions will be performed 3-5 days/week and will consist of walking for up to 60 minutes/day at 55% VO2max.
  Arms: Exercise - Continuous Walking

SUMMARY:
The purpose of this study is to assess whether 4-months of interval-walking exercise training improves glycemic control in individuals with type 2 diabetes mellitus. The effects of interval-walking training will be compared to continuous-walking exercise in a randomised, controlled trial design. Changes in glycemic control will be examined using oral glucose tolerance tests (OGTT) with stable isotope methodology. In addition, insulin sensitivity and secretion will be examined using glucose clamps combined with glucagon-like peptide 1 (GLP-1) and glucose-dependent insulinotropic polypeptide (GIP).

ELIGIBILITY:
Inclusion Criteria:

* age 18 to 80
* normal glucose tolerance, impaired glucose tolerance, or type 2 diabetes (as evidenced by use of oral hypoglycemic medication or 2-hour OGTT glucose > 11.1 mmol/l)

Exclusion Criteria:

* Insulin treatment or type 1 diabetes
* BMI <19 or >40
* Physically active
* Undergoing weight-loss/gain
* Pregnancy
* Contraindication to exercise (ECG/CPX)
* Significant cardiovascular disease
* History of renal/hepatic/gastrointestinal/pulmonary disease
* Clotting or bleeding disorders

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2010-08; Primary Completion 2012-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Glycemic Control | 0 and 4 months
  Fasting glucose, two-hour glucose during OGTT, and hemoglobin A1c will be measured.

SECONDARY OUTCOMES:
Beta-cell Function | 0 and 4 months
  Glucose tolerance tests and hyperglycemic clamps combined with GLP-1 / GIP will be conducted. Glucose tracer kinetics and C-peptide deconvolution will be used to assess pancreatic function.
Body Composition | 0 and 4 months
  DXA and MRI will be used to assess changes in whole body and regional adiposity.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas P Solomon, Ph.D., Principal Investigator — Rigshospitalet, Denmark; Kristian Karstoft, M.D., Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

REFERENCES:
- [Derived] Karstoft K, Winding K, Knudsen SH, James NG, Scheel MM, Olesen J, Holst JJ, Pedersen BK, Solomon TP. Mechanisms behind the superior effects of interval vs continuous training on glycaemic control in individuals with type 2 diabetes: a randomised controlled trial. Diabetologia. 2014 Oct;57(10):2081-93. doi: 10.1007/s00125-014-3334-5. Epub 2014 Aug 7. PMID 25099941
- [Derived] Solomon TP, Malin SK, Karstoft K, Kashyap SR, Haus JM, Kirwan JP. Pancreatic beta-cell function is a stronger predictor of changes in glycemic control after an aerobic exercise intervention than insulin sensitivity. J Clin Endocrinol Metab. 2013 Oct;98(10):4176-86. doi: 10.1210/jc.2013-2232. Epub 2013 Aug 21. PMID 23966244
- [Derived] Solomon TP, Malin SK, Karstoft K, Haus JM, Kirwan JP. The influence of hyperglycemia on the therapeutic effect of exercise on glycemic control in patients with type 2 diabetes mellitus. JAMA Intern Med. 2013 Oct 28;173(19):1834-6. doi: 10.1001/jamainternmed.2013.7783. No abstract available. PMID 23817567
- [Derived] Karstoft K, Winding K, Knudsen SH, Nielsen JS, Thomsen C, Pedersen BK, Solomon TP. The effects of free-living interval-walking training on glycemic control, body composition, and physical fitness in type 2 diabetic patients: a randomized, controlled trial. Diabetes Care. 2013 Feb;36(2):228-36. doi: 10.2337/dc12-0658. Epub 2012 Sep 21. PMID 23002086